CLINICAL TRIAL: NCT05928130
Title: Determining the Minimum Effective Volume of Plyometric Training for Inducing Changes in Lower Limb Strength, Power, and Muscle Electrical Activity During Functional Performance Testing in Sedentary Individuals
Brief Title: Efficiency in 4-week Plyometric Training: Lower Limb Improvement in Sedentary Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rodrigo Lizama Perez (Other)
Responsible Party: Sponsor-Investigator, Rodrigo Lizama Perez, secondary investigator, Universidad de Granada
Organization: Universidad de Granada (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IDAFISAD 64202
Record Dates: First submitted 2023-05-16; First posted 2023-07-03 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Plyometric Exercise; Sedentary Behavior
Keywords: Plyometric exercise; Lower extremity; Sedentary behavior; Muscle strength; Electromyography
MeSH Terms: conditions — Sedentary Behavior

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Volume Training Group (Experimental): Participants in this group will undergo a plyometric training protocol at a known effective volume that is expected to induce changes in lower limb strength, power, and muscle activity.
  Interventions: Other: plyometric training protocol
- Reduced Volume Training Group (Experimental): Participants in this group will undergo a plyometric training protocol at a lower volume than the Volume Training Group, aiming to determine if a lower volume still leads to significant improvements in lower limb strength, power, and muscle activity.
  Interventions: Other: plyometric training protocol
- Control Group (No Intervention): Participants in this group will not undergo any plyometric training and will serve as a comparison to assess the natural progression of lower limb strength, power, and muscle activity without intervention.

INTERVENTIONS:
Other: plyometric training protocol — The plyometric training program will last for 4 weeks, with three sessions per week. The plyometric exercises will be performed immediately after a warm-up. The program will incorporate bilateral, unilateral, acyclic, cyclic, horizontal, vertical, lateral, and diagonal movements involving both slow and fast movements.
  Each session will include 4-5 plyometric exercises, with 2-10 sets per exercise and 1-10 repetitions per set. The training volume will progressively increase from the 1st to the 2nd week and then the intensity will increase while the volume decreases from the 3rd to the 4th week in both intervention groups. However, the final volume will vary by 50% between the groups.
  Arms: Reduced Volume Training Group; Volume Training Group

SUMMARY:
The goal of this clinical trial is to compare the effects of different volumes of plyometric training on lower limb muscle strength, power, and muscle activity in sedentary individuals. The main question[s] it aims to answer are:

* What is the minimum volume of plyometric training that can induce changes in lower limb strength and power variables?
* How does muscle activity in the lower limbs vary with different volumes of plyometric training?

Participants will be asked to:

* Complete questionnaires to determine their level of physical activity.
* Attend pre and post-evaluations of lower limb muscle activity, strength, and power during an instrumented sit-to-stand test.
* Perform lower limb plyometric exercises, such as jumps, hops, and bounds.
* Attend supervised training sessions three times a week for a duration of 4 weeks.

Researchers will compare three groups to see if the minimum volume of plyometric training can be identified.

ELIGIBILITY:
Inclusion Criteria:

* Subjects without lower limb musculoskeletal injuries in the past six months.
* Without previous lower limb surgery in the past two years
* Being sedentary

Exclusion Criteria:

* Medical conditions that could compromise their participation (including cardiovascular disease).

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2023-07-30 (Actual); Primary Completion 2024-01-30 (Actual); Study Completion 2024-02-20 (Actual)

PRIMARY OUTCOMES:
Change from baseline muscle strength at 4 weeks | Baseline (pre-intervention), and two days after the last training session
  level of lower limb muscle strength during an instrumented sit to stand test
Change from baseline muscle power at 4 weeks | Baseline (pre-intervention), and two days after the last training session
  level of lower limb muscle power during an instrumented sit to stand test
Change from baseline muscle activity at 4 weeks | Baseline (pre-intervention), and two days after the last training session
  level of lower limb electromyographic activity during an instrumented sit to stand test

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad San Sebastián, sede Valdivia., Valdivia, Chile

IPD SHARING:
Plan to Share IPD: No